CLINICAL TRIAL: NCT00616746
Title: Interactive Psychopharmacologic Effects of Alcohol and Nicotine in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: 0607001614
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Alcohol Consumption; Tobacco Use
Keywords: Alcohol, nicotine
MeSH Terms: conditions — Alcohol Drinking; Tobacco Use | interventions — Nicotine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Three test days, within-subject design.
  Interventions: Drug: Nicotine; Drug: Ethanol

INTERVENTIONS:
Drug: Nicotine — 1.0 microg/kg/min IV x 10 minutes
Drug: Ethanol — IV

SUMMARY:
The purpose of this study is to characterize the interactive effects of acute intravenous (IV) alcohol and nicotine administration in male and female smokers and nonsmokers who use alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, 21 to 50 years old.

Exclusion Criteria:

* Alcohol or Nicotine Naive

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Behavioral and Cognitive Measures | Baseline and Test Day

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, M.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven Campus, West Haven, Connecticut, United States